CLINICAL TRIAL: NCT02561780
Title: Youth Mental Health Awareness Study and Early Intervention Research Project
Brief Title: Impact of a Mental Health Curriculum for High School Students on Knowledge and Stigma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Robert Milin, Associate Professor, Department of Psychiatry, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2010011
Record Dates: First submitted 2015-09-18; First posted 2015-09-28 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Mental Disorders; Education Curriculum; Comparative Effectiveness Research; Early Intervention; Adolescents
Keywords: Mental Health Knowledge; Stigma; Mental Health Literacy
MeSH Terms: conditions — Mental Disorders; Social Stigma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Curriculum (Active Comparator): The curriculum is a mental health literacy resource designed to inform high school curricula and contains six distinct modules: 1) stigma of mental illness; 2) understanding mental health and mental illness; 3) information on specific mental illnesses; 4) experiences of mental illness; 5) seeking help and finding support; and 6) the importance of positive mental health.
  A research assistant trained teachers on The Curriculum Guide content in a half-day session. Teachers implemented The Curriculum Guide, which requires approximately 6 hours of classroom time, during regular instruction of the Healthy Living course.
  Interventions: Behavioral: Curriculum
- Curriculum +eLearning Follow-up (Active Comparator): The curriculum is a mental health literacy resource designed to inform high school curricula and contains six distinct modules: 1) stigma of mental illness; 2) understanding mental health and mental illness; 3) information on specific mental illnesses; 4) experiences of mental illness; 5) seeking help and finding support; and 6) the importance of positive mental health.
  A research assistant trained teachers on The Curriculum Guide content in a half-day session. Teachers implemented The Curriculum Guide, which requires approximately 6 hours of classroom time, during regular instruction of the Healthy Living course. Students are asked to complete follow-up modules online. These modules are only accessible after completion of the Healthy Living course.
  Interventions: Behavioral: Curriculum; Behavioral: eLearning Follow-up
- Teaching As Usual (Control) (No Intervention): Schools randomized to this arm of the study received the unadulterated Healthy Living course, taught as usual.

INTERVENTIONS:
Behavioral: Curriculum — A mental health educational resource delivered in the classroom by trained educators
  Other Names: The Curriculum Guide
  Arms: Curriculum; Curriculum +eLearning Follow-up
Behavioral: eLearning Follow-up — An online mental health education module that students access individually
  Other Names: online follow-up learning module
  Arms: Curriculum +eLearning Follow-up

SUMMARY:
This study examines the effectiveness of a school based mental health literacy intervention for high school students, on improving mental health knowledge and reducing stigma. Twenty-four high schools in the regional area of Ottawa, Canada were randomly assigned to either the curriculum or control condition at a two to one ratio. The educational curriculum was integrated within grade 11 and 12 Provincial "Healthy Living" courses, delivered by teachers, and replaced existing educational content on mental health.

DETAILED DESCRIPTION:
There is limited evidence and consensus on the effectiveness of school-based mental health educational programs, and no standardization for mental health education being taught in schools. This study examines the effectiveness of a school-based mental health literacy intervention for adolescents, on knowledge and stigma. A secondary objective was to determine the generalizability and applicability of an educational resource for mental health in high schools.

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled in the Healthy Living course of participating Ottawa area community high schools.

Exclusion Criteria:

* Students not enrolled in the Healthy Living course of participating Ottawa area community high schools.
* Students with an English reading and comprehension level lower than the sixth grade

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 534 (Actual)
Dates: Start 2011-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Self-Report Knowledge of Mental Illness Scale | Immediately following completed delivery of The Curriculum Guide
  15 multiple choice questions about mental illness computed to provide a total score of mental health knowledge for each participant
Self-Report Attitudes Towards Mental Illness Scale | Immediately following completed delivery of The Curriculum Guide
  A Likert scale of 8 statements about characteristics of individuals with mental illness computed to provide a total score of positive attitudes towards mental illness for each participant

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Milin, MD, Principal Investigator — Associate Professor

REFERENCES:
- [Derived] Milin R, Kutcher S, Lewis SP, Walker S, Wei Y, Ferrill N, Armstrong MA. Impact of a Mental Health Curriculum on Knowledge and Stigma Among High School Students: A Randomized Controlled Trial. J Am Acad Child Adolesc Psychiatry. 2016 May;55(5):383-391.e1. doi: 10.1016/j.jaac.2016.02.018. Epub 2016 Mar 8. PMID 27126852